CLINICAL TRIAL: NCT04912973
Title: Clinical & Biomechanical Outcome After Robotic Total Knee Arthroplasty by Comparing Inverse Kinematic Alignment and Mechanical Alignment - Gait Analysis and Performance Testing
Brief Title: Assessment With Gait Analysis of Robotic Total Knee Arthroplasty Using Inverse Kinematic Alignment
Acronym: RATKA-CBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philip Winnock de Grave, MD (Other)
Collaborators: AZ Delta (Other)
Responsible Party: Sponsor-Investigator, Philip Winnock de Grave, MD, Principal Investigator, AZ Delta
Organization: AZ Delta (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3222020000151
Record Dates: First submitted 2021-05-17; First posted 2021-06-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee arthroplasty; robotic surgery; alignment; inverse kinematic alignment; mechanical alignment; gait analysis; performance testing
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- inverse Kinematic Alignment (Active Comparator)
  Interventions: Procedure: Robotically Assisted Total Knee Arthroplasty - Knee Replacement
- adjusted Mechanical Alignment (Active Comparator)
  Interventions: Procedure: Robotically Assisted Total Knee Arthroplasty - Knee Replacement

INTERVENTIONS:
Procedure: Robotically Assisted Total Knee Arthroplasty - Knee Replacement — Robotically Assisted Total Knee Arthroplasty with a particular alignment strategy
  Other Names: Triathlon Total Knee System of Stryker with Mako Robotic Platform; Triathlon Total Knee Replacement of Stryker

SUMMARY:
Postoperative function and patient satisfaction are becoming increasingly relevant in patients after knee arthroplasty surgery. Despite adequate preoperative planning, improved surgical techniques and rehabilitation protocols, only 75%-85% of patients seems satisfied after TKA procedurs. Implant positioning and component alignment are determining factors in patient outcome. Currently, different alignment strategies in TKA surgery are used such as Mechanical Alignment (MA) and Kinematical Alignment (KA). Recently, a new and individualized alignment strategy (inverse Kinematic Alignment/iKA) was introduced. Preliminary 1-year results of iKA are promising, however, clinical and functional outcome on the medium and longterm should be investigated. This project aims to compare patients with iKA TKA with MA TKA on clinical, functional and biomechanical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. Received a primary total knee replacement (incl. patella) robotically-assisted
3. Male or female
4. Age between 50 and 80
5. Able to walk independently

Exclusion Criteria:

1. Revision surgery
2. Patient with a history of neurological, psychiatric or neurodegenerative disease
3. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
4. Other musculoskeletal lesions that may affect the gait pattern

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Gait Analysis - walking speed - faster is better | 2 year
  Spatio Temporal Parameters are captured with infra-red camera during gait: velocity
Performance Testing - step-up step-down speed - faster is better | 2 year
  Spatio Temporal Parameters are captured with infra-red camera during functional movements: velocity

SECONDARY OUTCOMES:
Patient Reported Outcome Measures - Oxford Knee Score (OKS): maximum score (best) is 48/48; worst score is 0/48 | baseline - 1 year - 2 year
  Questionnaire - Oxford Knee Score

CONTACTS AND LOCATIONS:
Locations (1):
- AZDelta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No